CLINICAL TRIAL: NCT06487546
Title: Repletion of Ergothioneine in Patients With Kidney Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tammy Lisa Sirich, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 75743
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Esrd
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Ergothioneine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ergothioneine (Experimental): Ergothioneine (range 5 mg to 25 mg) oral daily for up to 16 weeks
  Interventions: Dietary Supplement: Ergothioneine

INTERVENTIONS:
Dietary Supplement: Ergothioneine — This is a 1-arm study in which participants will take ergothioneine daily with dose range of 5 mg to 25 mg daily. Blood levels of ergothioneine will be monitored while taking daily ergothioneine and after ergothioneine is stopped.

SUMMARY:
Dialysis removes potentially harmful chemicals from the blood but can also remove potentially valuable chemicals. One potentially valuable chemical called ergothioneine, which comes from the diet, is low in the blood of people receiving dialysis. For this research study, the investigators hope to learn how well a daily ergothioneine supplement will replenish the levels in the blood of people with kidney failure.

ELIGIBILITY:
Inclusion Criteria:

* kidney failure receiving hemodialysis or peritoneal dialysis

Exclusion Criteria:

* blood transfusion within 90 days
* taking supplements which contain ergothioneine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
erythrocyte levels of ergothioneine | weeks 1, 2, 4, 8, 12, and 16 (while taking ergothioneine); and weeks 20 and 24 (after stopping ergothioneine)
  ergothioneine levels will be measured in whole blood
plasma levels of ergothioneine | weeks 1, 2, 4, 8, 12, and 16 (while taking ergothioneine); and weeks 20 and 24 (after stopping ergothioneine)
  ergothioneine levels will be measured in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Veterans Affairs Palo Alto, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halliwell B, Tang RMY, Cheah IK. Diet-Derived Antioxidants: The Special Case of Ergothioneine. Annu Rev Food Sci Technol. 2023 Mar 27;14:323-345. doi: 10.1146/annurev-food-060822-122236. Epub 2023 Jan 9. PMID 36623925
- [Background] Chen L, Zhang L, Ye X, Deng Z, Zhao C. Ergothioneine and its congeners: anti-ageing mechanisms and pharmacophore biosynthesis. Protein Cell. 2024 Feb 29;15(3):191-206. doi: 10.1093/procel/pwad048. PMID 37561026